CLINICAL TRIAL: NCT03161626
Title: A Multicenter, Post-Marketing Registry Study of COAGADEX® in the Peri-operative Management of Patients With Moderate or Severe Hereditary Factor X Deficiency Undergoing Major Surgery
Brief Title: Registry Study of COAGADEX® Patients With Moderate or Severe Hereditary Factor X Deficiency Undergoing Major Surgery
Status: Completed | Type: Observational
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Other Study IDs: Ten06
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Factor 10 Deficiency
MeSH Terms: conditions — Factor X Deficiency | interventions — Factor X

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate to Severe Factor X Deficiency
  Interventions: Drug: Coagadex

INTERVENTIONS:
Drug: Coagadex — Plasma-driven blood coagulation factor X concentration
  Other Names: Factor X

SUMMARY:
This is a non-interventional, multicenter, post-marketing registry study in three patients with moderate or severe hereditary FX deficiency, to assess Coagadex administered peri-operatively for hemostatic cover in major surgery during routine post-marketing use.

DETAILED DESCRIPTION:
The primary objective is to collect additional surgical data on the clinical effectiveness of Coagadex, in a post-marketing environment, for peri-operative hemostatic cover during major surgery in patients with moderate or severe hereditary factor X (FX) deficiency.

The secondary objective is to review safety data on Coagadex through the collection of any Adverse Drug Reactions (ADRs) from the first dose of Coagadex in the hospital prior to the surgical procedure until the first follow-up after discharge (i.e., follow-up completed) and Serious ADRs up until the post-operative care follow-up has been completed. Data on any deaths and pregnancies reported within this time period will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients >12 years of age with severe or moderate hereditary FX deficiency. Severe is defined as <1 IU/dL and moderate as 1 to 5 IU/dL (3)
* Patients who have given written informed consent (for sites in the USA this will include the Health Insurance Portability and Accountability Act (HIPAA) authorization statement), OR, in the case of 12-18 year olds, written informed consent from the parents/ guardians and where appropriate assent from the child
* Patients requiring major surgery. Major surgery is defined as procedures typically requiring:

  * full anesthesia or regional anesthesia, e.g. epidural or spinal and
  * involving the opening of major cavities such as thoracic, abdominal surgery; orthopedic surgery, and Caesarean section (C-section) and
  * requiring at least one overnight stay in hospital (16)

Exclusion Criteria:

* Patients known to be pregnant, unless the surgery is C-section.
* Patients who participated in a clinical study trial in the last 30 days prior to study enrolment, except if they have been involved in another study involving Coagadex.
* Patients with a known history of inhibitor development to FX.
* Patients who are required or expected to take other factor X-containing medications during or after surgery.
* Patients with existing known thrombocytopenia (platelets < 50 x 109/L).
* Patients with existing known clinically significant renal disease (creatinine >200 µmol/L).
* Patients with existing known clinically significant liver disease (ALT levels greater than three times the upper limit of normal).
* Patients with existing known other coagulopathy or thrombophilia.
* Patients with a known intolerance or allergy to Coagadex or its excipients.
* Patients known to have abused chemicals or drugs within the past 12 months.
* Patients with a history of unreliability or non-cooperation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate or severe hereditary Factor X deficiency undergoing major surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Retrospective surgical data collection | 12 months
  Blood loss (mL)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Florida Health, Gainesville, Florida
  - Tulane University Hospitals and Clinics, New Orleans, Louisiana
  - West Michigan Cancer Center, Kalamazoo, Michigan